CLINICAL TRIAL: NCT07029373
Title: A Prospective Clinical Study for Analyzing Plasma Calcitonin Gene-Related Peptide (CGRP) Levels in Patients With Head and Neck Malignancies Undergoing Radiotherapy
Brief Title: Plasma Calcitonin Gene-Related Peptide (CGRP) Levels in Patients With Head and Neck Malignancies Undergoing Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Other Study IDs: 2025-989
Record Dates: First submitted 2025-06-01; First posted 2025-06-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; Radiotherapy-related pain; Calcitonin gene-related peptide
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prospective observational study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective study investigates the dynamic changes in plasma calcitonin gene-related peptide (CGRP) levels during radiotherapy and their association with radiotherapy-related pain in patients with head and neck malignancies.

DETAILED DESCRIPTION:
Radiotherapy-related pain is a major clinical challenge that significantly affects the long-term quality of life and treatment adherence of patients with head and neck cancer. Current analgesic strategies offer limited efficacy, and reliable biomarkers for predicting pain risk are lacking. In recent years, calcitonin gene-related peptide (CGRP) has drawn increasing attention for its critical role in chronic pain regulation, as demonstrated in various pain models. However, no systematic studies have yet investigated the expression patterns and clinical relevance of CGRP in radiotherapy-induced pain among patients with head and neck malignancies. This single-center, prospective observational study aims to enroll patients with head and neck cancer receiving either definitive or postoperative adjuvant radiotherapy. Plasma samples will be collected before, during, and after radiotherapy for measurement of CGRP levels. Pain intensity will be simultaneously assessed using the Numeric Rating Scale (NRS) and the Brief Pain Inventory-Short Form (BPI-SF). The study seeks to explore the dynamic changes in plasma CGRP levels throughout the radiotherapy course and to analyze their correlation with patient-reported pain, thereby providing potential insights into biomarker-based pain prediction and management strategies in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Histologically confirmed head and neck malignancy

Planned to receive definitive or postoperative adjuvant radiotherapy

Radiotherapy duration ≥ 4 weeks, with irradiation field involving the oral cavity, pharynx, or neck region

Able and willing to provide written informed consent

Able to complete pain assessments and blood sample collection

Exclusion Criteria:

* History of significant chronic pain prior to radiotherapy (e.g., postherpetic neuralgia, rheumatoid arthritis)

Presence of uncontrolled hypertension, diabetes, or migraines

Presence of other active malignancies or major systemic diseases (e.g., severe hepatic or renal dysfunction)

Currently receiving or recently received treatments that may significantly affect pain perception (e.g., opioids, antidepressants)

Pregnant or breastfeeding

Inability to complete follow-up or poor treatment compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with histologically confirmed head and neck malignancies scheduled to receive definitive or postoperative adjuvant radiotherapy (≥4 weeks) involving the oral cavity, pharynx, or neck will be enrolled. Exclusion criteria include pre-existing significant chronic pain (e.g., postherpetic neuralgia, rheumatoid arthritis), uncontrolled hypertension, diabetes, or migraines, other active malignancies or major systemic diseases (e.g., severe hepatic/renal dysfunction), recent or current use of medications affecting pain perception (e.g., opioids, antidepressants), pregnancy or breastfeeding, and inability to complete follow-up or poor treatment compliance.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma CGRP level | Baseline (prior to the initiation of radiotherapy), At the end of the third week of radiotherapy (approximately 21±2 days after the 15th radiotherapy session), Within one week after the completion of radiotherapy.
  To assess dynamic changes in CGRP levels during the course of radiotherapy.
Correlation between CGRP levels and pain scores (NRS and BPI-SF) | Baseline (prior to the initiation of radiotherapy), At the end of the third week of radiotherapy (approximately 21±2 days after the 15th radiotherapy session), Within one week after the completion of radiotherapy.
  To evaluate the association between CGRP expression and radiotherapy-induced pain.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — Department of Biotherapy, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China